CLINICAL TRIAL: NCT00430209
Title: Neurovascular Coupling in Eyes of Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 083-GUK-2006-001; Swiss National Foundation (Other Grant/Funding Number: 3200B0-113685)
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
We hypothesize that glaucoma patients demonstrate an impaired retinal vascular response to the flicker stimulus, and that this disturbance is predictive of the progression of glaucomatous damage.

The response of a major temporal superior and inferior retinal artery and vein to a 60 seconds 12.5 Hz flicker light stimulation in 50 glaucoma patients, 50 ocular hypertensives and 50 controls (using the Retinal Vessel Analyzer) and to investigate how intraocular pressure relates to neurovascular coupling. In addition, 50 glaucoma patients and 50 ocular hypertension patients will be followed for 3 years for functional (visual field, automated perimetry with Octopus device) and morphological (retinal nerve fiber layer thickness, Optical Coherence Tomography Stratus ocular coherence tomography (OCT) device) glaucomatous damage progression, in order to test the predictive power of the retinal vascular flicker response for glaucoma progression.

DETAILED DESCRIPTION:
Rationale: The term neurovascular coupling refers to the vascular response to an increased neuronal activity. The contact of the nerve terminals to the cortical blood vessels is mostly realized through astrocytes. A major defining property of glaucoma, cupping of the optic disc, implies tissue remodeling of the optic nerve head and involves an astrocytic responses. A malfunction of the astrocytes in glaucoma may lead not only to the hallmark of glaucoma, cupping and death of retinal ganglion cells, but also to an accompanying or even preceding disturbance in ocular neurovascular coupling. The retinal vascular bed was chosen because of the high reproducibility of the dynamic retinal vessel diameter analysis and because recently the hypoxia-inducible factor 1α was found not only in the glia of the optic nerve head but also in the retina of glaucomatous donor eyes and predominantly in retinal locations closely concordant with the locations of visual field defects recorded in these eyes, raising questions about the site of primary damage in glaucoma. It is hoped that this research project will help provide a workable tool and a model able not only to identify a risk factor for glaucoma, but in the future to explore possible therapeutic avenues to modify the course of the disease.

Working hypothesis: We hypothesize that glaucoma patients demonstrate an impaired retinal vascular response to the flicker stimulus, and that this disturbance is predictive of the progression of glaucomatous damage

Subjects and Methods The present protocol intends to explore the response of a major temporal superior and inferior retinal artery and vein to a 60 seconds 12.5 Hz flicker light stimulation in 50 glaucoma patients, 50 ocular hypertensives and 50 controls (using the Retinal Vessel Analyzer) and to investigate how intraocular pressure relates to neurovascular coupling. In addition, 50 glaucoma patients and 50 ocular hypertension patients will be followed for 3 years for functional (visual field, automated perimetry with Octopus device) and morphological (retinal nerve fiber layer thickness, Optical Coherence Tomography Stratus OCT device) glaucomatous damage progression, in order to test the predictive power of the retinal vascular flicker response for glaucoma progression. Patients will be recruited in the University Eye Clinic Basel, a notification in the University Hospital of Basel and/or advertisement in a newspaper will inform potential healthy volunteers of the opportunity to participate in a scientific research project.

Study Course: Study is divided in the cross-sectional and in the cohort part. In the former, first the screening examination will be performed, to establish an eligibility of a patient / control subject for the study. Thereafter, the measurements described above will follow, which will conclude the cross-sectional part of the study. Glaucoma patients and patients with ocular hypertension will be offered a possibility to enter the cohort-study, with a 3-year follow-up embedded in the clinical routine and consisting of biannual repeated measurements outlined above.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma
* ocular hypertension

Exclusion Criteria:

* highest ever measured intraocular pressure (IOP) equal or higher than 30 mmHg
* peripapillary hemorrhage
* any suspicion of progression
* PEX (pseudo exfoliations syndrome) or pigment dispersion syndrome
* a history of an acute glaucoma attack
* chamber angle dysgenesia
* any form of secondary glaucoma
* diabetes
* high levels of blood lipids
* systemic or ocular circulatory diseases
* medication, drugs, alcohol, smoking
* systolic blood pressure above 145mmHg or a diastolic above 95mmHg
* visual acuity worse than 20/25
* high ametropia (spherical equivalent < -5 diopters or > +3 diopters)
* astigmatism above 2 diopters
* significant cataract
* filtering procedures

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma patients ocular hypertensives normal controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response to flicker light in glaucoma | up to 3 years
  Response to flicker light in glaucoma, ocular hypertension (OHT) and normal subjects

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Eye Clinic, Basel
Locations (1):
- University Eye Clinic, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Gugleta K, Waldmann N, Polunina A, Kochkorov A, Katamay R, Flammer J, Orgul S. Retinal neurovascular coupling in patients with glaucoma and ocular hypertension and its association with the level of glaucomatous damage. Graefes Arch Clin Exp Ophthalmol. 2013 Jun;251(6):1577-85. doi: 10.1007/s00417-013-2276-9. Epub 2013 Feb 19. PMID 23417339
- [Derived] Gugleta K, Kochkorov A, Waldmann N, Polunina A, Katamay R, Flammer J, Orgul S. Dynamics of retinal vessel response to flicker light in glaucoma patients and ocular hypertensives. Graefes Arch Clin Exp Ophthalmol. 2012 Apr;250(4):589-94. doi: 10.1007/s00417-011-1842-2. Epub 2011 Oct 19. PMID 22008947
- [Derived] Portmann N, Gugleta K, Kochkorov A, Polunina A, Flammer J, Orgul S. Choroidal blood flow response to isometric exercise in glaucoma patients and patients with ocular hypertension. Invest Ophthalmol Vis Sci. 2011 Sep 9;52(10):7068-73. doi: 10.1167/iovs.11-7758. PMID 21828157